CLINICAL TRIAL: NCT02904642
Title: Randomized Controlled Trial of the Impact of Mobile Phone Delivered Reminders and Unconditional Travel Subsidies on Measles Vaccination in Western Kenya: The Mobile and Scalable Innovations for Measles Immunization (M-SIMI) Trial
Brief Title: Mobile and Scalable Innovations for Measles Immunization: a Randomized Controlled Trial
Acronym: M-SIMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Kenya Medical Research Institute (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Dustin Gibson, Assistant Scientist, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KEMRI SERU-3311
Record Dates: First submitted 2016-09-08; First posted 2016-09-19 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Measles
Keywords: SMS reminder; incentive; mobile phone; Immunization
MeSH Terms: conditions — Measles

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): All enrolled caregivers will receive a congratulatory text message at enrollment which indicates who is conducting the study and which also includes a general-health related saying, "The greatest wealth is health". No additional text messages or travel subsidies will be sent to caregivers randomized to the control arm.
- SMS reminder (Experimental): At enrollment, participants will be told to expect 2 SMS reminders for measles vaccine; first, at 3 days before and second, on the day before the scheduled measles vaccine at 9 months of age. At most, enrolled caregivers will receive three text messages (two for the measles vaccine and one for welcoming mother to the study). Text messages will be sent in English, Kiswahili or Dholuo language, according to the mother's preference. These reminders will have information about the child's scheduled immunization date.
  Interventions: Behavioral: SMS reminder
- SMS reminder + Unconditional Incentive (Experimental): Participants will receive SMS reminders as described in the SMS reminder arm. Additionally, participants will be sent a 150 Kenyan Shillings (KES) incentive to the mobile phone number they provided at enrollment. The incentive will be delivered three days before the child turns nine months (i.e. sent on the same day as the first SMS reminder). Caregivers will receive the mobile-money incentive unconditionally. The intent of the incentive is to help offset the costs associated with transportation to the clinic. The transaction costs associated with mobile-money transactions will be borne by the study such that mothers will receive the full 150 KES.
  Interventions: Behavioral: SMS reminder; Behavioral: Unconditional Incentive

INTERVENTIONS:
Behavioral: SMS reminder — Caregivers will receive two text message reminders for their child's measles immunization scheduled for 9 months of age
  Arms: SMS reminder; SMS reminder + Unconditional Incentive
Behavioral: Unconditional Incentive — A mobile-money incentive in the amount of 150 Kenyan Shillings will be transferred to the enrolled caregiver's mobile phone when the child reaches nine months of age
  Arms: SMS reminder + Unconditional Incentive

SUMMARY:
The overall objective is to test the impact of short message service (SMS) reminders, with or without unconditionally provided mobile-money incentives, can improve measles vaccination coverage in rural western Kenyan infants.

DETAILED DESCRIPTION:
Primary Objective The primary objective is to determine if text message reminders, with or without unconditionally provided incentives, can increase the proportion of children who receive measles vaccination by 15% at age ten months as compared to control arm children.

Secondary Objectives

1. To conduct a secondary analysis of the primary outcome using survival analysis and time-to-immunization curves.
2. To determine if there is a differential effect on measles vaccine coverage based on mobile phone ownership and distance to the clinic.
3. To examine the effect of the interventions on measles coverage measured at twelve months of age.
4. To examine the completeness and costs of identifying children through a CHW approach versus the standard HDSS approach.
5. To evaluate the effect of the interventions on coverage of second dose of measles vaccine at 24 months. This secondary objective is contingent on receiving additional funding.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver of infant aged 6-8 months at time of enrollment
* Self-reported resident of one of the study villages; where the definition of a resident is defined by caregiver
* Willing to sign informed consent for the study

Exclusion Criteria:

* Child of enrolled caregiver has already received one dose of measles vaccine, not including any supplemental measles vaccines
* Caregiver plans to move away in the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 537 (Estimated)
Dates: Start 2016-12-06 (Actual); Primary Completion 2017-04-04 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
Measles vaccination coverage | 10 months
  Proportion of children receiving measles vaccination by 10 months of age by study arm

SECONDARY OUTCOMES:
Time to measles vaccination (in days) using Kaplan-Meier Survival Analysis | 12 months
  As a secondary analysis of the primary outcome, time-to-measles immunization curves will be constructed using the Kaplan-Meier method and study arms will be compared using the Cox model. The 25th, 50th, and 75th percentiles for time to immunization and the number of days delayed, in relation to the measles due date, will also be reported for each vaccine and by study arm.
Proportion of children who receive measles vaccination stratified by demographic variables | 10 months
  A priori we will conduct sub group analyses of the primary outcome for mobile phone ownership, birth order of the enrolled caregiver's child, and time to clinic. Additional variables for subgroup analyses will come from a risk factor analysis of not receiving measles vaccination in the control arm
Measles vaccination coverage at 12 months | 12 months
  Proportion of children who receive measles vaccination by twelve months of age by study arm
Vaccination coverage for second dose of measles vaccine at 24 months. | 24 months
  This outcome is dependent on receiving more funding

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kagucia EW, Ochieng B, Were J, Hayford K, Obor D, O'Brien KL, Gibson DG. Impact of mobile phone delivered reminders and unconditional incentives on measles-containing vaccine timeliness and coverage: a randomised controlled trial in western Kenya. BMJ Glob Health. 2021 Jan;6(1):e003357. doi: 10.1136/bmjgh-2020-003357. PMID 33509838
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276
- [Derived] Gibson DG, Kagucia EW, Were J, Obor D, Hayford K, Ochieng B. Text Message Reminders and Unconditional Monetary Incentives to Improve Measles Vaccination in Western Kenya: Study Protocol for the Mobile and Scalable Innovations for Measles Immunization Randomized Controlled Trial. JMIR Res Protoc. 2019 Jul 9;8(7):e13221. doi: 10.2196/13221. PMID 31290405